CLINICAL TRIAL: NCT02803944
Title: Long Term Effects of Azithromycin in Patients With Cystic Fibrosis Using the National Database
Brief Title: Continuous Azithromycin in Cystic Fibrosis Patients Beyond Two Years
Acronym: AZITHRO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0240
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
Keywords: azithromycin; cystic fibrosis; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis | interventions — Azithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic fibrosis patients taking azithromycin: Cystic fibrosis patients taking azithromycin continuously for two years.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
Azithromycin is an antibiotic currently prescribed continuously in cystic fibrosis patients. It was shown that this treatment taken every day or every week for 12 months, can improve the respiratory state of patients. From the second year of treatment, it would appear there is more profit to continue such treatment.

The main objective is to study the association between continuous use of azithromycin and lung function measured by Forced expiratory volume in one second (FEV1), after two years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cystic Fibrosis (whatever the genetic form)
* Age ≥ 8 years
* FEV ≥ 30% the year of azithromycin (N0)
* Continuous treatment with azithromycin for at least 2 years.

Exclusion Criteria:

-

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eligible population consists of patients over 7 years old with CF followed in Resource Centres and Competence for Cystic Fibrosis (CRCM) France.
Sampling Method: Non-Probability Sample
Enrollment: 2055 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1). | yearly recorded, 2 years before initiation of Azithromycin and 4 years after initiation of Azithromycin

SECONDARY OUTCOMES:
Body Mass Index (BMI) | yearly recorded, 2 years before initiation of Azithromycin and 4 years after initiation of Azithromycin
Number of IV antibiotics cures | yearly recorded, 2 years before initiation of Azithromycin and 4 years after initiation of Azithromycin
Pseudomonas aeruginosa colonization | yearly recorded, 2 years before initiation of Azithromycin and 4 years after initiation of Azithromycin

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle DURIEU, Pr, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France